CLINICAL TRIAL: NCT03551197
Title: Impact of Exercise on Lung Function in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Change of Lung Function After Exercise in Patients With Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-HXNK-001
Record Dates: First submitted 2018-05-09; First posted 2018-06-11 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Exercise; Lung Function Decreased; Quality of Life
Keywords: Pulmonary Disease, Chronic Obstructive; exercise; lung function; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Respiratory Insufficiency | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: There is only one group.Patients with diagnosis of Chronic Obstructive Pulmonary Disease are recruited.Subjects will be examined at baseline and after 3 months' treatment of budesonide and formoterol.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Budesonide and formoterol bid (Experimental): At baseline,lung function test,blood oxygen saturation and pulse are measured before and after 6-min walk test for each subject.Quality of life is assessed through questionnaires including modified Medical Research Council dyspnoea scale(mMRC),St George's Respiratory Questionnaire(SGRQ),clinical chronic obstructive pulmonary questionnaire(CCQ) and chronic obstructive pulmonary disease assessment test(CAT).And then budesonide(160ug) and formoterol(4.5ug) bid will be given to the subjects for 3 months.The subjects will have a follow-up visit with all the examinations mentioned above after 3 months' treatment.
  Interventions: Drug: Budesonide and formoterol bid

INTERVENTIONS:
Drug: Budesonide and formoterol bid — At baseline,lung function test,blood oxygen saturation and pulse are measured before and after 6-min walk test for each subject.Quality of life is assessed through questionnaires including modified Medical Research Council dyspnoea scale(mMRC),St George's Respiratory Questionnaire(SGRQ),clinical chronic obstructive pulmonary questionnaire(CCQ) and chronic obstructive pulmonary disease assessment test(CAT).And then budesonide(160ug) and formoterol(4.5ug) bid will be given to the subjects for 3 months.The subjects will have a follow-up visit with all the examinations mentioned above after 3 months' treatment.
  Other Names: SYMBICORT TURBUHALER

SUMMARY:
The purpose of this study is to evaluate the changes of lung function before and after the exercise in patients with chronic obstructive pulmonary disease.The assessment of quality of life is also carried out through questionnaires.

DETAILED DESCRIPTION:
This is a randomized,open-label study to research the changes of lung function before and after exercise in patients with chronic obstructive pulmonary disease .At baseline,lung function test,blood oxygen saturation and pulse are measured before and after 6-min walk test for each subject.Quality of life is assessed through questionnaires including modified Medical Research Council dyspnoea scale(mMRC),St George's Respiratory Questionnaire(SGRQ),Clinical Chronic Obstructive Pulmonary Questionnaire(CCQ) and chronic obstructive pulmonary assessment test(CAT).And then budesonide(160ug) and formoterol(4.5ug) bid will be given to the subjects for 3 months.The subjects will have a follow-up visit with all the examinations mentioned above after 3 months' treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 to 80 years-old, inclusive.
* A clinical diagnosis of chronic obstructive pulmonary disease according to the Global Initiative for Chronic Obstructive Disease(GOLD 2018) guidelines.
* Post bronchodilator (following inhalation of salbutamol) forced expired volume in one second(FEV1)/forced vital capacity(FVC) ratio ≤0.70.
* Willing and able to provide written informed consent.
* Willing and able to attend all study visits and adhere to all study assessments and procedures.

Exclusion Criteria:

* Severe comorbidities including unstable cardiac or pulmonary disease or any other medical conditions including unstable ischemic heart disease,unstable cardiac arrhythmia or heart failure,life threatening arrhythmias,etc.
* Recent history of chronic obstructive pulmonary disease exacerbation requiring hospitalization or need for increased treatments for chronic obstructive pulmonary disease within 6 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-13 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Changes of forced expired volume in one second(FEV1) after 6-min walk test compared with resting state | At resting state and after 6-min walk test
  Forced expired volume in one second(FEV1) is measured by Jaeger MasterScreen Pulmonary Function Test System before and after 6-min walk test.

SECONDARY OUTCOMES:
Changes of inspiratory capacity(IC) after 6-min walk test compared with resting state | At resting state and after 6-min walk test
  Inspiratory capacity(IC) is measured by Jaeger MasterScreen Pulmonary Function Test System before and after 6-min walk test.
Changes of blood oxygen saturation after 6-min walk test compared with resting state | At resting state and after 6-min walk test
  Blood oxygen saturation is measured before and after 6-min walk test.
Changes of pulse after 6-min walk test compared with resting state | At resting state and after 6-min walk test
  Pulse is measured before and after 6-min walk test.
Changes of forced expired volume in one second(FEV1) after 3 months' treatment compared with baseline | Change from baseline to 3 months
  At baseline,forced expired volume in one second(FEV1) is measured.After 3 months's treatment of budesonide and formoterol,FEV1 will be measured again.
Changes of inspiratory capacity(IC) after 3 months' treatment compared with baseline | Change from baseline to 3 months
  At baseline,inspiratory capacity(IC) is measured.After 3 months's treatment of budesonide and formoterol,IC will be measured again.
Changes of diffusion function after 3 months' treatment compared with baseline | Change from baseline to 3 months
  At baseline,diffusion function is measured.After 3 months's treatment of budesonide and formoterol,diffusion function will be measured again.
Changes of impulse forced oscillometry parameters after 3 months' treatment compared with baseline | Change from baseline to 3 months
  At baseline,impulse forced oscillometry parameters are measured.After 3 months's treatment of budesonide and formoterol,impulse forced oscillometry parameters will be measured again.
Changes of modified Medical Research Council dyspnoea scale(mMRC) scores after 3 months' treatment compared with baseline | Change from baseline to 3 months
  At baseline,quality of life is assessed by modified Medical Research Council dyspnoea scale(mMRC).After 3 months's treatment of budesonide and formoterol,the mMRC scores will be measured again.
Changes of St George's Respiratory Questionnaire(SGRQ) scores after 3 months' treatment compared with baseline | Change from baseline to 3 months
  At baseline,quality of life is assessed by St George's Respiratory Questionnaire(SGRQ).After 3 months's treatment of budesonide and formoterol,the SGRQ scores will be measured again.
Changes of clinical chronic obstructive pulmonary questionnaire(CCQ) scores after 3 months' treatment compared with baseline | Change from baseline to 3 months
  At baseline,quality of life is assessed by clinical chronic obstructive pulmonary disease questionnaire(CCQ).After 3 months's treatment of budesonide and formoterol,the scores will be measured again.
Changes of chronic obstructive pulmonary disease assessment test(CAT) scores after 3 months' treatment compared with baseline | Change from baseline to 3 months
  At baseline,quality of life is assessed by chronic obstructive pulmonary disease assessment test(CAT).After 3 months's treatment of budesonide and formoterol,the test will be performed again.
The distance and steps of 6-min walk test | Change from baseline to 3 months
  Both the the distance and steps are measured

CONTACTS AND LOCATIONS:
Overall Officials: Huapeng Yu, Principal Investigator — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China